CLINICAL TRIAL: NCT02288650
Title: Incidence of Post-operative Vomitings (POV) After Early Refeeding in Pediatric Day Case Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 5547
Record Dates: First submitted 2013-07-25; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Post-operative Vomiting Incidence; Pediatric Day Case Surgery

ARMS (2):
- Liberal group (Experimental): Early refeeding
  Interventions: Other: early refeeding
- Control group (Sham Comparator): Refeeding in the day case ward (usual practice)
  Interventions: Other: refeeding only in the recovery room (usual practice).

INTERVENTIONS:
Other: early refeeding
  Arms: Liberal group
Other: refeeding only in the recovery room (usual practice).
  Arms: Control group

SUMMARY:
At the child, the post-operative vomitings (POV) remain the main post-operative complication in term of frequency. They also represent the first cause of unforeseen hospitalization in day case surgery. The causes of POV are multiple, including in particular the post-operative prescription of opioids. The role of the premature refeeding remains discussed.

Up to the age of 4 years, acute pain is difficult to distinguish from other causes of distress (anxiety, anger but also hunger) being able to make prescribe wrongly opioids in post-operative.

The main objective of this study is to estimate the POV in pediatric day case surgery after early refeeding with clear liquids in the recovery room or only in the day case wards (usual practice).

The secondary objectives are to estimate the time on returning to the day case ward, at home, the post-operative opioid consumption, early refeeding adverse effects (desaturation, swallowing trouble)

ELIGIBILITY:
Inclusion Criteria:

* Patient of less than 4 years old
* A pediatric day case surgery scheduled

Exclusion Criteria:

* Child lower age or 3 month old equal
* Premature child of conceptional age lower than 60 weeks
* Anesthetic or surgical constraint dissuading day case surgery or early refeeding
* Digestive pathology predisposing to the VPO (Hernia hiatal, gastro-oesophageal reflux)
* treatment interfering with emesis (imidazoles, neuroleptic)
* Period of exclusion defined by another study

Ages: 3 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 808 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Time between withdrawal of orotracheal tube and POV | The participant are followed for 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Derived] Chauvin C, Schalber-Geyer AS, Lefebvre F, Bopp C, Carrenard G, Marcoux L, Mayer JF, Schwaab C, Joshi GP, Diemunsch P. Early postoperative oral fluid intake in paediatric day case surgery influences the need for opioids and postoperative vomiting: a controlled randomized trialdagger. Br J Anaesth. 2017 Mar 1;118(3):407-414. doi: 10.1093/bja/aew463. PMID 28203729